CLINICAL TRIAL: NCT02599987
Title: Effectiveness of Inspiratory Muscle Training in Respiratory Muscle Strength, Chest Wall Volume, Diaphragm Thickness and Mobility in Patients With End-stage Renal Disease: Randomized Clinical Trial
Brief Title: Inspiratory Muscle Training in Patients With End-stage Renal Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, ANA IRENE CARLOS DE MEDEIROS, Principal Investigator, Universidade Federal de Pernambuco
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 48538315.4.0000.5208
Record Dates: First submitted 2015-11-04; First posted 2015-11-09 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2017-01

CONDITIONS: Kidney Disease
MeSH Terms: conditions — Kidney Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Inspiratory Muscle Training Group (Experimental): Will use the breathing coach POWERbreathe® Classic Light. Participants will hold the workout three sets of 30 inspirations, 2 sessions per day, 7 days per week for 8 weeks. The training group will carry with IMT load of 50% of MIP. Weekly, patients attend the Cardiopulmonary Physical Therapy Laboratory for evaluation of MIP and load adjustment, performing a training session in the presence of the therapist, while other sessions will be held by the participant at home and registered in the diary training. The training took place with the patient sitting in chair with a back, with knees and hips flexed to 90 °, the participant will use a nose clip and the device coupled to the nozzle mouth, will be instructed to diaphragmatic breathing pattern.
  Interventions: Device: POWERbreathe® Classic Light
- Sham Group (Sham Comparator): Will use the breathing coach POWERbreathe® Classic Light. Participants will hold the workout three sets of 30 inspirations, 2 sessions per day, 7 days per week for 8 weeks. The sham group will carry without load, but will be subjected to the same procedures in the experimental group (simulation of load adjustment in the Cardiopulmonary Physical Therapy Laboratory) to ensure blinding of the study, other sessions will be held by the participant at home and registered in the diary training. The training took place with the patient sitting in chair with a back, with knees and hips flexed to 90 °, the participant will use a nose clip and the device coupled to the nozzle mouth, will be instructed to diaphragmatic breathing pattern.
  Interventions: Device: POWERbreathe® Classic Light

INTERVENTIONS:
Device: POWERbreathe® Classic Light — Inspiratory Muscle Training

SUMMARY:
Background: Patients with chronic kidney disease on hemodialysis may have reduced diffusion capacity, lung function and gas exchange due to mechanical and hemodynamic changes in the respiratory system, and decreased respiratory muscle strength resulting from uremic myopathy. The inspiratory muscle training (IMT) appears as an instrument to improve the inspiratory muscle strength, with positive effects on functional capacity and quality of life of kidney patients, however, the effects of IMT were not addressed in the specific variables of the respiratory system and to date there are no studies on the use of daily training in this population. Objective: To evaluate the effectiveness of daily inspiratory muscle training on respiratory muscle strength, chest wall volume, diaphragm thickness and mobility of end-stage renal disease patients. Methods: A randomized controlled clinical trial to be developed in Cardiopulmonary Physical Therapy Laboratory of the Universidade Federal de Pernambuco (UFPE) during the period from November 2015 to December 2016. The sample is composed of 24 individuals aged 18 and 65, having CKD, to perform hemodialysis for at least twelve months and provide inspiratory muscle weakness. Patients will be divided into two groups, the training group will be IMT with POWER-breathe®, load of 50% of MIP, duration of three sets of 30 inspirations, frequency of two sessions per day, 7 days a week for 8 weeks, since the sham group will be subjected to the same procedure (duration and frequency), but without load. Participants will be assessed before and after intervention through a global assessment form, questionnaire Kidney Disease Quality of Life Instrument Short Form - KDQOL-SF, diaphragmatic ultrasound, opto-electronic plethysmography, spirometry, manometer and six-minute walk test.

ELIGIBILITY:
Inclusion Criteria:

* Have a chronic kidney disease
* Hemodialysis for a minimum period of twelve months
* Inspiratory muscle weakness, with MIP <80cmH2O for men and <60cmH2O for women

Exclusion Criteria:

* Neurological deficit
* Chronic lung disease
* Severe heart disease (unstable angina and acute myocardial infarction)
* Decompensated diabetes
* Infectious disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-11; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Respiratory muscle strength | 2 months
  Evaluate by manometer
Diaphragm thickness | 2 months
  Evaluate by ultrasound

SECONDARY OUTCOMES:
Chest wall volume | 2 months
  Evaluate by opto-electronic plethysmography
Pulmonary function | 2 months
  Evaluate by Spirometry
Walking distance | 2 months
  Evaluate by six-minute walk test
Quality of life | 2 months
  Evaluate by questionnaire Kidney Disease Quality of Life Instrument Short Form - KDQOL-SF
Diaphragm mobility | 2 months
  Evaluate by ultrasound

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiopulmonary Physiotherapy Laboratory of UFPE, Recife, Pernambuco, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Caruso P, Albuquerque AL, Santana PV, Cardenas LZ, Ferreira JG, Prina E, Trevizan PF, Pereira MC, Iamonti V, Pletsch R, Macchione MC, Carvalho CR. Diagnostic methods to assess inspiratory and expiratory muscle strength. J Bras Pneumol. 2015 Mar-Apr;41(2):110-23. doi: 10.1590/S1806-37132015000004474. PMID 25972965
- [Background] Pellizzaro CO, Thome FS, Veronese FV. Effect of peripheral and respiratory muscle training on the functional capacity of hemodialysis patients. Ren Fail. 2013;35(2):189-97. doi: 10.3109/0886022X.2012.745727. Epub 2012 Nov 30. PMID 23199095
- [Background] Pessoa IM, Houri Neto M, Montemezzo D, Silva LA, Andrade AD, Parreira VF. Predictive equations for respiratory muscle strength according to international and Brazilian guidelines. Braz J Phys Ther. 2014 Sep-Oct;18(5):410-8. doi: 10.1590/bjpt-rbf.2014.0044. Epub 2014 Sep 12. PMID 25372003
- [Background] Figueiredo RR, Castro AA, Napoleone FM, Faray L, de Paula Junior AR, Osorio RA. Respiratory biofeedback accuracy in chronic renal failure patients: a method comparison. Clin Rehabil. 2012 Aug;26(8):724-32. doi: 10.1177/0269215511431088. Epub 2012 Jan 18. PMID 22257505
- [Background] Enright SJ, Unnithan VB, Heward C, Withnall L, Davies DH. Effect of high-intensity inspiratory muscle training on lung volumes, diaphragm thickness, and exercise capacity in subjects who are healthy. Phys Ther. 2006 Mar;86(3):345-54. PMID 16506871
- [Background] Aliverti A, Pedotti A. Opto-electronic plethysmography. Monaldi Arch Chest Dis. 2003 Jan-Mar;59(1):12-6. PMID 14533277
- [Background] ATS Committee on Proficiency Standards for Clinical Pulmonary Function Laboratories. ATS statement: guidelines for the six-minute walk test. Am J Respir Crit Care Med. 2002 Jul 1;166(1):111-7. doi: 10.1164/ajrccm.166.1.at1102. No abstract available. PMID 12091180
- [Background] Duarte PS, Ciconelli RM, Sesso R. Cultural adaptation and validation of the "Kidney Disease and Quality of Life--Short Form (KDQOL-SF 1.3)" in Brazil. Braz J Med Biol Res. 2005 Feb;38(2):261-70. doi: 10.1590/s0100-879x2005000200015. Epub 2005 Feb 15. PMID 15785838
- [Derived] Medeiros AIC, Brandao DC, Souza RJP, Fuzari HKB, Barros CESR, Barbosa JBN, Leite JC, Cavalcanti FCB, Dornelas de Andrade A, de Melo Marinho PE. Effects of daily inspiratory muscle training on respiratory muscle strength and chest wall regional volumes in haemodialysis patients: a randomised clinical trial. Disabil Rehabil. 2019 Dec;41(26):3173-3180. doi: 10.1080/09638288.2018.1485181. Epub 2018 Jul 27. PMID 30052475